CLINICAL TRIAL: NCT03170687
Title: Comparative Outcomes Between Foot Cast and Short Leg Cast in the Patients With Acute Closed Fracture of Proximal Fifth Metatarsal (Zone II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jatupon Kongtharvonskul (Other)
Collaborators: Police General Hospital (Other)
Responsible Party: Sponsor-Investigator, Jatupon Kongtharvonskul, clinical doctor in section of clinical epidermiology and biostatistic, Ramathibodi Hospital
Organization: Ramathibodi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53/2560
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Acute Closed Fracture of Proximal Fifth Metatarsal (Zone II)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot cast (Experimental)
  Interventions: Device: short foot cast
- short leg cast (Active Comparator)
  Interventions: Device: short leg cast

INTERVENTIONS:
Device: short foot cast — metatarsal foot cast
  Arms: foot cast
Device: short leg cast — full short leg cast
  Arms: short leg cast

SUMMARY:
This study aims to compare outcomes of short leg cast and foot cast for treatment acute fifth metatarsal fracture (Zone II).

DETAILED DESCRIPTION:
A randomized controlled trial will conducts between January 2017 and January 2019, participants with acute fifth metatarsal fracture (Zone II) will recruit for this study at the orthopedic outpatient clinic of a police general hospital, Bangkok, Thailand. A total of 100 patients will randomly allocate to receive foot cast or short leg cast. acute closed fracture of proximal fifth metatarsal (zone II) patients.

ELIGIBILITY:
Inclusion Criteria:acute closed fracture of proximal fifth metatarsal (zone II) with following criteria

1. History of trauma and pain at lateral side of foot
2. Tenderness at base of 5th metatarsal
3. Radiographic finding shown fracture line at proximal 5th metatarsal bone

Exclusion Criteria:

1. more than 1 week
2. comminuted or multiple fracture
3. Open fracture
4. Ligament and tendon injury
5. Previous injury complication: nonunion, delayed union
6. Malignancy
7. refuse to inform consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
VAS | 8 weeks
  visual analog score

SECONDARY OUTCOMES:
AOFAS | 8 weeks
  foot score
union rate | 8 weeks
  radiographic union
complication | 8 weeks
  skin ulcer or compartment syndrome

OTHER OUTCOMES:
rescue medication | 8 weeks
  paracetamol or NSAIDs

CONTACTS AND LOCATIONS:
Locations (1):
- Jatupon Kongtharvonskul, Bangkok, Select..., Thailand

IPD SHARING:
Plan to Share IPD: No